CLINICAL TRIAL: NCT00473096
Title: Assessing the Efficacy of a CDSS for Breast Cancer
Brief Title: Efficacy Study of an Educational Program for Decision Support for Breast Cancer
Acronym: H-6019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Maria Jibaja Weiss, Associate Professor, Duncan Cancer Center, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DAMD17-98-1-8022
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Breast Neoplasms
Keywords: Decision making; Patient Education; Indigency; Minority group
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Informed breast cancer surgical treatment

SUMMARY:
The purpose of this study is to develop and test an informative computer-based program to help women in making good choices among options for treating early stage breast cancer. Women who are exposed to the computerized program will, when compared to women who receive standard of care offered at the hospital: (a) be more knowledgeable about treatment options,(b) be more satisfied with their treatment decision, and (c) be more assured about their treatment choice.

DETAILED DESCRIPTION:
The purpose of this project is to develop and test a computer-based decision support system on breast cancer for low-income women who speak English or Spanish. This project is designed to respond to the under utilization of breast conserving surgery by women with early stage breast cancer, as indicated by both national and local data on treatment choices. The literature suggests that underuse of BCS by women for whom it is the recommended therapy may relate to inadequacies in efforts to educate them about treatment options. The program was designed to convey information to women with varying levels of reading ability. This was done through multimedia approaches which include voice-over narrative in simple English or Spanish, and use of photo novella and/or "soap opera" presentation of situational material that allows women to explore possible consequences associated with different decisions.

Comparison(s): Women exposed to the computer-based decision support program on breast cancer treatment, receiving standard care and education offered at two public hospitals, compared to women exposed to standard care and education at the same public hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Breast cancer diagnosis in stages I, IIA, IIB, or IIIA
* Candidates for surgery
* Speak English or Spanish

Exclusion Criteria:

* Breast cancer diagnosis in stages 0, IIIB, or IV
* Recurrent breast cancer or inflammatory breast carcinoma
* Not eligible for lumpectomy with radiation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Treatment decisions more consistent with preferences (utilities)at pre-operation
Breast cancer treatment knowledge at 6 month and 1 year
Certainty about treatment choice at pre-operation

SECONDARY OUTCOMES:
Satisfaction with decision at the pre-operation, 6 month and 1 year
Preferences for decision making at pre-operation
Satisfaction with the decision making process at pre-operation, 6 month and 1 year
Functional status at 6 month and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Jibaja Weiss, EdD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Result] Jibaja-Weiss ML, Volk RJ, Friedman LC, Granchi TS, Neff NE, Spann SJ, Robinson EK, Aoki N, Robert Beck J. Preliminary testing of a just-in-time, user-defined values clarification exercise to aid lower literate women in making informed breast cancer treatment decisions. Health Expect. 2006 Sep;9(3):218-31. doi: 10.1111/j.1369-7625.2006.00386.x. PMID 16911136
- [Result] Jibaja-Weiss ML, Volk RJ, Granch TS, Nefe NE, Spann SJ, Aoki N, Robinson EK, Freidman LC, Beck JR. Entertainment education for informed breast cancer treatment decisions in low-literate women: development and initial evaluation of a patient decision aid. J Cancer Educ. 2006 Fall;21(3):133-9. doi: 10.1207/s15430154jce2103_8. PMID 17371175